CLINICAL TRIAL: NCT04238897
Title: A Prospective Randomized Control Study to Evaluate the Effect of Ticon Aspherical Daily Disposable Soft Contact Lens on Myopia Control
Brief Title: To Evaluate the Efficacy and Safety of Aspherical Soft Contact Lens in Myopia Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: APP Vision Care Inc. (Industry)
Collaborators: National Taiwan University Hospital (Other); Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1011128M
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Myopia
Keywords: myopia control; soft contact lens; eye diseases
MeSH Terms: conditions — Myopia; Eye Diseases | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Intervention Model Description: paired-eye design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticon Aspherical Daily Disposable Soft Contact Lens (Experimental): The subject will be requested to wear lens 8 hours a day, 5 days a week at least. The contact lens will be worn and replaced every day. All subjects will be followed for 1 year post device allocation with a brief clinical assessment at 1 day, 1 week, 1, 3, 6, 9, 12 months.
  Interventions: Device: soft contact lens
- Ticon Daily Soft Contact Lens (Placebo Comparator): The subject will be requested to wear lens 8 hours a day, 5 days a week at least. The contact lens will be worn and replaced every day. All subjects will be followed for 1 year post device allocation with a brief clinical assessment at 1 day, 1 week, 1, 3, 6, 9, 12 months.
  Interventions: Device: soft contact lens

INTERVENTIONS:
Device: soft contact lens

SUMMARY:
The objective of this study is to demonstrate that the Ticon Aspherical Daily Disposable Soft Contact Lens could retard myopia progress in youth

DETAILED DESCRIPTION:
This study is designed as a prospective, multicenter, randomized, double blinded, controlled, paired-eye comparison study. At least 60 evaluable subjects with myopia progression ≧ 0.75 D in the past 12 months will be recruited from 2 study sites. The experimental soft contact lens with aspherical design (Ticon Aspherical) will be randomly assigned to either the right eye or the left eye of the subject , then the fellow eye will be assigned a control lens with a single vision distance (SVD) soft contact lens (Ticon). Both lenses will be worn at least 8 hours a day, 5 days a week for 1 year. All lenses will be replaced every day. Brief assessment of the clinical findings will be followed up for one year at 1 day, 1 week, 1, 3, 6, 9, 12 months upon allocation. The primary efficacy outcome is change in spherical equivalent refraction (SER) measured by cycloplegic autorefraction over 12 months. The secondary outcome is change in axial eye length (AXL) measured over 12 months. The secondary outcome measure is used to corroborate any changes in SER

ELIGIBILITY:
Inclusion Criteria:

* Myopia (SE) between -1.00D to -8.00D
* Astigmatism less than or equal to 1.75D
* Myopia progression ≧0.75 D in the past 12 months
* Best Corrected Visual Acuity (BCVA): 0.9 Snellen or better
* Willingness to wear contact lens constantly
* Availability for follow-up for at least 1 year
* Parent's understanding and acceptance
* have an acceptable surrogate capable of giving legally authorized consent on behalf of the subject

Exclusion Criteria:

* Anisometropia greater than 2.00D
* Presence of ocular disease preventing wear of contact lens
* Severe ocular or systemic allergies
* Taking any medication that might have an impact on contact lens wear or that might influence the outcome of the clinical trial
* Ocular or systemic condition that might affect refractive development
* Atropine/Pirenzepine treatment for myopia control in the past 1 month
* Prior use of Ortho-K lenses
* Dry eye with Schimer Test (basal secretion test) < 5mm/5min or other physical condition that would contraindicate contact lens wear

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Spherical Equivalent Refraction (SER) | 12 months
  The change in spherical equivalent refraction (SER) measured by cycloplegic autorefraction over 12 months.

SECONDARY OUTCOMES:
Axial Eye Length (AXL) | 12 months
  The change in axial eye length (AXL) measured over 12 months. Axial length is measured after cycloplegia using optical biometry.

OTHER OUTCOMES:
Primary safety Endpoints | 12 months
  All dispensed eyes over all follow-up visits. Measured on a scale of 0-4 with 0=no findings and 4=severe findings. Epithelial edema, epithelial microcysts, corneal staining, limbal & bulbar injection, conjunctival abnormalities, corneal neovascularization and infiltrates will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Hsun Tsai, M.D., Study Chair — National Taiwan University Hospital; Elizabeth P Shen, M.D., Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation; Hsiao-Sang Chu, M.D., Principal Investigator — National Taiwan University Hospital; Han-Chih Cheng, M.D., Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation

REFERENCES:
- [Derived] Shen EP, Chu HS, Cheng HC, Tsai TH. Center-for-Near Extended-Depth-of-Focus Soft Contact Lens for Myopia Control in Children: 1-Year Results of a Randomized Controlled Trial. Ophthalmol Ther. 2022 Aug;11(4):1577-1588. doi: 10.1007/s40123-022-00536-5. Epub 2022 Jun 23. PMID 35737291